CLINICAL TRIAL: NCT00325026
Title: Randomized Trial Comparing Misoprostol and Foley Bulb for Labor Induction in the Preterm Gestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 594-2004
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Premature Birth; Cervical Ripening
Keywords: Preterm gestation; Cervical ripening; Labor induction; Misoprostol; Foley bulb
MeSH Terms: conditions — Premature Birth | interventions — Misoprostol

INTERVENTIONS:
Drug: Misoprostol
Device: Foley bulb

SUMMARY:
The purpose of this study is to compare the time to delivery of two different cervical ripening methods on the preterm gestation.

DETAILED DESCRIPTION:
Labor induction for the preterm gestation is indicated for various maternal and fetal indications. The preterm cervix, however, is frequently not favorable for induction. Multiple methods have been evaluated in the term gestation. As these comparison studies have not included the preterm gestation, this study seeks to evaluate these two methods in terms of safety, efficacy and time to delivery.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation, gestational age 23-35 weeks, indication for induction

Exclusion Criteria:

* multiple gestation, non-cephalic presentation, previous uterine surgery, rupture of membranes, intrauterine fetal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time to vaginal delivery

SECONDARY OUTCOMES:
Rate of chorioamnionitis
Incidence of abnormal fetal heart rate tracings
Rate of postpartum hemorrhage
Incidence of NICU admissions

CONTACTS AND LOCATIONS:
Overall Officials: Keri a Baacke, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264